CLINICAL TRIAL: NCT06993272
Title: Relaxation Music for Patients With Chronic Pain From IBS, Crohn's, or Colitis
Brief Title: Relaxation Music for Chronic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sean D Young, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5116
Record Dates: First submitted 2025-04-18; First posted 2025-05-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: IBS - Irritable Bowel Syndrome; IBD - Inflammatory Bowel Disease
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MIndful Jazz (Experimental): Participants in this group will watch an introduction to jazz appreciation and mindfulness training video, including the use of jazz for pain tolerance prior to the 4-week intervention. Participants in the Mindful Jazz Group will be informed that listening to music they are not comfortable with (i.e., jazz) can enhance long-term pain tolerance.
  Interventions: Behavioral: MIndful Jazz
- Reggae Stereotypes (Experimental): Reggae Stereotype Group: Participants in this group will be told about he stereotype of reggae in making people more calm. They will listen to reggae music over the 4 weeks.
  Interventions: Behavioral: Reggae Stereotypes
- Traditional Mindfulness (Experimental): Participants in this group will listen to a traditional mindfulness practice over the 4 weeks
  Interventions: Behavioral: Traditional Mindfulness
- Pain Psychoeducation (Active Comparator): Participants listen to the same playlist each week of the 4-weeks. It's an audio recording of the pain psychoeducation video they watch during training. Video: https://www.youtube.com/watch?v=azwEQXh5enA
  Interventions: Behavioral: Pain psychoeducation

INTERVENTIONS:
Behavioral: MIndful Jazz — Mindful Jazz Group: Participants in this group will watch an introduction to jazz appreciation and mindfulness training video, including the use of jazz for pain tolerance prior to the 4-week intervention. Participants in the Mindful Jazz Group will be informed that listening to music they are not comfortable with (i.e., jazz) can enhance long-term pain tolerance.
  Arms: MIndful Jazz
Behavioral: Reggae Stereotypes — Reggae Stereotype Group: Participants in this group will be told about he stereotype of reggae in making people more calm. They will listen to reggae music over the 4 weeks.
  Arms: Reggae Stereotypes
Behavioral: Traditional Mindfulness — Participants will listen to a traditional mindfulness practice over the 4 weeks
  Arms: Traditional Mindfulness
Behavioral: Pain psychoeducation — Participants listen to an audio recording of the pain psychoeducation video they watch during training over the 4 weeks. Video: https://www.youtube.com/watch?v=azwEQXh5enA
  Arms: Pain Psychoeducation

SUMMARY:
Chronic pain is a common complaint in inflammatory bowel disease (IBD). Compounding these concerns, opioid analgesics are frequently used to treat severe acute pain. An estimated 30% of chronic pain patients due to IBD report opioid use. Those who continue to use opioids can develop opioid misuse, and opioid misuse portends addiction and overdose so there is a need for better, non-addictive treatment options.

Music interventions effectively reduce pain and pain-related symptomology. Meta-analytic results indicate listening to music can reduce acute and chronic pain. Music listening also decreases emotional distress from pain as well as the use of pain medication. Music interventions have demonstrated these positive effects on pain across a number of settings, including surgical, in-patient, and community settings. Importantly, due to the ubiquity of music - especially freely available online music - music interventions are easily accessible and highly scalable.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Living in U.S.
* Have a pain rating related to IBS, Crohn's, or Colitis of five or greater in average pain on a 0-10 numeric rating scale in the preceding week
* Have had pain related to IBS, Crohn's, or Colitis for at least 3 months and for at least 15 days in the preceding 30 days
* GAD Score (Moderate to Severe Anxiety)

Exclusion Criteria:

* Are currently using or have used prescription opioids in the past 3 months
* Have a current cancer diagnosis
* In one of our prior music studies
* Have formal experience with mindfulness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain, Enjoyment, General Activity Scale (PEG) | Baseline and 4 weeks
  Pain Intensity:
  Measure: The PEG scale will be used to assess the magnitude of pain sensations experienced by participants in the past week.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No